CLINICAL TRIAL: NCT01259947
Title: Chemical Composition and Therapeutic Effects of Lippia Alba (Mill.) N. E. Brown Leaves Ethanolic Extract in Patients With Migraine
Brief Title: Lippia Alba for Migraine Prophylaxis and Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fabio Carmona (Other)
Responsible Party: Sponsor-Investigator, Fabio Carmona, Technical coordinator, Casa Espirita Terra de Ismael
Organization: Casa Espirita Terra de Ismael (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LALBA201012
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Migraine Disorders
Keywords: headache; migraine; medicinal plant; essential oil; phytotherapy
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lippia alba (Experimental)
  Interventions: Drug: Lippia alba (Mill.) N. E. Brown ethanolic extract

INTERVENTIONS:
Drug: Lippia alba (Mill.) N. E. Brown ethanolic extract — 1-2 drops per kilogram per day, PO, twice a day

SUMMARY:
Abstract Background: There is no universally accepted and effective prophylaxis of migraine headache episodes. Thus the investigators aimed to investigate the effects of Lippia alba (Mill.) N. E. Brown, an herb with many effects on central nervous system, on pain frequency and intensity of migraine patients.

Methods: Patients were enrolled in a prospective, phase 2, non-controlled cohort study to orally receive ethanolic extract of L. alba leaves (1-2 drips/kg/day). Headache intensity and frequency of episodes were recorded before and after 30-60 days of treatment. The investigators also studied the chemical composition of its essential oil by gas chromatography-mass spectrometry.

Results: The investigators described for the first time a particular L. alba chemotype with geranial and carvenone as major compounds. With treatment, both frequency and intensity of pain episodes significantly decreased from baseline to first reassessment date. More than 80% of patients experienced a minimum 50% reduction on pain intensity and frequency. No side effects were reported.

Conclusions: Treatment with a geranial plus carvenone chemotype of L. alba ethanolic extract is a cheap, widely available, highly effective therapy to reduce both the intensity and the frequency of headache episodes of migraine patients with no side effects.

Keywords: headache, migraine, medicinal plant, essential oil, phytotherapy

ELIGIBILITY:
Inclusion Criteria:

* Migraine diagnostic

Exclusion Criteria:

* Patient's request

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-07; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul Conde, MD, Principal Investigator — Reserva EcoCerrado Brasil; Ana MS Pereira, PhD, Study Chair — Casa Espirita Terra de Ismael
Locations (1):
- Naturoterapia Sinho Mariano, Araxá, Minas Gerais, Brazil

REFERENCES:
- [Derived] Carmona F, Angelucci MA, Sales DS, Chiaratti TM, Honorato FB, Bianchi RV, Pereira AM. Lippia alba (Mill.) N. E. Brown hydroethanolic extract of the leaves is effective in the treatment of migraine in women. Phytomedicine. 2013 Jul 15;20(10):947-50. doi: 10.1016/j.phymed.2013.03.017. Epub 2013 Apr 30. PMID 23639189
- [Derived] Conde R, Correa VS, Carmona F, Contini SH, Pereira AM. Chemical composition and therapeutic effects of Lippia alba (Mill.) N. E. Brown leaves hydro-alcoholic extract in patients with migraine. Phytomedicine. 2011 Nov 15;18(14):1197-201. doi: 10.1016/j.phymed.2011.06.016. Epub 2011 Jul 29. PMID 21802924